CLINICAL TRIAL: NCT06236516
Title: One Fraction Simulation-Free Treatment With CT-Guided Stereotactic Adaptive Radiotherapy for Patients With Oligometastatic and Primary Lung Tumors (ONE STOP)
Brief Title: One Fraction Simulation-Free Treatment With CT-Guided Stereotactic Adaptive Radiotherapy for Patients With Oligometastatic and Primary Lung Tumors
Acronym: ONE STOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202401015
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer; Oligometastatic Lung Tumor
Keywords: SBRT; Lung cancer; Oligometastatic cancer; Image-guided radiotherapy; Adaptive radiotherapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- One Fraction SBRT (Experimental): Consenting and eligible patients will receive a prescription dose of 25-34 Gy in one fraction with adaptation based on daily anatomic changes as per clinical standard of care.
  Interventions: Radiation: One fraction stereotactic body radiotherapy; Device: HyperSight; Device: Ethos

INTERVENTIONS:
Radiation: One fraction stereotactic body radiotherapy — Radiotherapy will consist of one-fraction SBRT using the Ethos linear accelerator and online adaptive treatment planning system.
  Other Names: SBRT
Device: HyperSight — HyperSight is a novel on-board imaging platform equipped with rapid-acquisition high-quality CBCT imager capable of acquiring images sufficient for both simulation and treatment.
Device: Ethos — Ethos is a unique ring-gantry CT-guided linear accelerator notable for having a dedicated artificial intelligence treatment planning system to allow for online adaptive radiotherapy.

SUMMARY:
Stereotactic body radiotherapy (SBRT) has become a standard of care for medically inoperable or high-risk operable early-stage non-small cell lung cancer (NSCLC) patients. It is also increasingly used to treat lung metastases in patients with oligometastatic disease. While SBRT is a powerful tool for the treatment of lung tumors, access to specialized treatment can be limited for patients who live far away from a treatment center. Geographic accessibility can be limiting even for patients receiving one fraction lung SBRT, as the typical consult, CT simulation, and one-fraction treatment workflow is typically at least two to three weeks from start to finish, with a minimum of three in-person appointments.

In this study, a high-quality cone beam CT (CBCT) on-board imaging platform (HyperSight; Varian Medical Systems, Palo Alto, CA) will be coupled with advanced motion management and treatment techniques as well as Ethos (Varian Medical Systems, Palo Alto, CA) daily online adaptation to simulation-free workflow for one fraction SBRT. This has the potential to reduce the time it takes a patient to be cured of their lung tumor from two to three weeks to two to three hours. In this novel workflow, patients will undergo telephone/online consent followed by a diagnostic scan-based pre-plan for one fraction SBRT. On the morning of treatment, a brief follow-up appointment will be followed by treatment on the HyperSight/Ethos platform. Patients will be treated using a simulation-free workflow. A HyperSight Thorax Slow protocol CBCT will be acquired for study purposes, and then the patient will be treated with online adaptive CBCT-guided radiotherapy on the Ethos/HyperSight platform. Treatment delivery will take place following contouring and treatment planning. Patients will undergo standard of care simulation imaging in parallel for comparison.

The purpose of this study is to evaluate the feasibility of a ONE fraction Simulation-free Treatment with CT-guided stereotactic adaptive radiotherapy for Oligometastatic and Primary lung tumors (ONE STOP) workflow for patients with small, peripheral primary or oligometastatic lung tumors.

ELIGIBILITY:
Inclusion Criteria:

* One of the following diagnoses:

  * Histologically or radiographically diagnosed stage I-IIA (AJCC, 8th ed.) non-small cell lung cancer .

    * Clinical AJCC stage I defined as stage 1A1 (T1a1N0M0, T1a tumor less than or equal to 1 cm), stage 1A2 (T1bN0M0, T1b tumor between 1 and 2 cm), and stage 1A3 (T1cN0M0, T1c tumor between 2 and 3 cm).
    * Clinical AJCC stage IB defined as T2aN0M0, T2a tumor between 3 and 4 cm.
    * Clinical AJCC stage IIA defined as T2bN0M0, T2b tumor between 4 and 5 cm.
  * Oligometastatic lung tumor secondary to a primary cancer of any type/histology. Oligometastatic patients may include patients with:

    * 1-5 sites of metastatic disease with at least one lung lesion intended to be treated with SBRT
    * More than 5 sites of metastatic disease with oligo-progressive disease in the lung intended to be treated with SBRT.
* Lesions must be small and peripheral.

  * Small is defined as max tumor dimension of 5 cm or less.
  * Peripheral is defined as greater than 2 cm from the proximal bronchial tree/mediastinum.
* Tumors and anatomy amenable to one-fraction lung SBRT confirmed by meeting of one-fraction lung SBRT target and constraint metrics on a diagnostic-scan based preplan.

  * Patients who do not meet this criterion will be screen fails and triaged to the standard lung SBRT workflow and treated off trial.
* Lesions must have a maximum superior to inferior motion of 1 cm on 4D-CT imaging.

  * Patients who do not meet this criteria will be screen fails and triaged to the standard lung SBRT workflow and treated off trial.
* At least 18 years of age.
* Able to understand and willing to sign an IRB approved written informed consent.

Exclusion Criteria:

* Past history of radiotherapy within the projected treatment field of any of the disease sites to be treated by ONE STOP SBRT.
* Pregnant and/or breastfeeding. Patient must have a negative pregnancy test within 14 days of ONE STOP SBRT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of the ONE STOP workflow | Day 1
  Feasibility is defined as the successful completion of the ONE STOP workflow through treatment delivery in at least 70% of patients.
  Successful completion of the workflow is defined as ONE STOP plan creation and delivery of the fraction using the study workflow in one on-table attempt.
  Unsuccessful completion of the workflow is defined as multiple attempts of the ONE STOP workflow for one patient without treatment delivery such that the study workflow is abandoned and a traditional one-, three-, or five-fraction plan is delivered.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Samson, M.D., MPHS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu